CLINICAL TRIAL: NCT05665556
Title: REgistry of Pulmonary Arterial Hypertension Associated With CONNECTIVE Tissue Diseases (RECONNECTIVE) at the National Institute of Medical Sciences and Nutrition Salvador Zubirán
Brief Title: REgistry of Pulmonary Arterial Hypertension Associated With CONNECTIVE Tissue Diseases (RECONNECTIVE)
Acronym: RECONNECTIVE
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Jose Luis Hernandez Oropeza, Head of the Pulmonary Hypertension Clinic, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: 3278
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Arterial Hypertension; Connective Tissue Diseases
Keywords: Pulmonary Arterial Hypertension; Connective Tissue Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Arterial Hypertension (Group I): Group I Pulmonary Arterial Hypertension associated with Connective Tissue Diseases
- Pulmonary Arterial Hypertension (Group IV): Group IV Pulmonary Arterial Hypertension associated with Connective Tissue Diseases

SUMMARY:
The RECONNECTIVE Registry is an observational single center study, focused on the subgroup of precapillary pulmonary hypertension related to connective tissue diseases. All patients will have hemodynamic confirmation by right heart catheterization and will be follow-up for at least 5 years from admission. All patients diagnosed with Group I Pulmonary Arterial Hypertension (PAH) associated with Connective Tissue Diseases (CTD) and Group IV Pulmonary Hypertension (PH) with CTD will be included. The purpose of the registry is to learn and understand the clinical outcomes and natural history of the pulmonary arterial hypertension in this subgroup of patients to improve the medical care and treatment.

DETAILED DESCRIPTION:
Connective tissue diseases represents an important risk factor for pulmonary hypertension, either due to vasculopathy or chronic pulmonary thromboembolism. These chronic conditions are characterized by being disabling, progressive and fatal in a short time and are caused by multiple mechanisms that results in remodeling of the pulmonary microvasculature and right heart failure.

In recent years, due to international registries, we have acquired a better understanding of high-risk subpopulations, their poor prognostic factors, and the results of specific combination therapies. In Mexico, the National Institute of Medical Sciences and Nutrition Salvador Zubirán (INCMNSZ) is a referral center for connective tissue diseases and pathologies of the pulmonary circulation. The RECONNECTIVE registry is a five years follow-up cohort that offers the possibility to obtain data regarding to the clinical characteristics and hemodynamic assesment of pulmonary circulation. The main objective is to evaluate the clinical course of the PAH in this subgroup of patients and their specific therapy for PAH.

ELIGIBILITY:
Inclusion Criteria:

* Incident and prevalent patients diagnosed with Group I associated with Connective Tissue Diseases (CTD)
* Incident and prevalent patients diagnosed with Group IV Pulmonary Arterial Hypertension (PAH) associated with Connective Tissue Diseases (CTD) with evidence of a chronic thromboembolic pulmonary disease by ventilation/perfusion pulmonary gammagraph or computed tomography pulmonary angiogram with at least three months of total anticoagulation therapy.
* Patient diagnosed with a connective tissue disease according to the classification criteria of the American College of Rheumatology.
* Precapillary pulmonary hypertension confirmed by right heart catheterization (RHC): Mean pulmonary arterial pressure (mPAP) >20 mm Hg with a pulmonary arterial wedge pressure ≤ 15 mm Hg and Pulmonary vascular resistance (PVR) ≥ 2.0 Wood units

Exclusion Criteria:

* Patients who meet the criteria for another group of pulmonary hypertension (Groups II, III or V).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Group I Pulmonary Arterial Hypertension (PAH) associated to Connective Tissue Diseases (CTD) and Group IV Pulmonary Hypertension group (PH) with CTD.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the clinical clinical course of Pulmonary Arterial Hypertension (PAH) associated with Connective Tissue Diseases (CTD) in a register of Mexican patients from the first visit and at every 6 months. | 5 years
  Outcome measure: Clinical worsening: defined internationally by death, lung or heart-lung transplantation, atrial septostomy, hospitalization due to worsening PAH, initiation of new PAH approved therapy, or worsening WHO functional class.

SECONDARY OUTCOMES:
World Health Organization functional class (I-IV) | 5 years
  Assesment of the functional class according to the World Health Organization (WHO) functional class (in scale from I-IV) in each scheduled visit (every 3 to 6 months) in the pulmonary hypertension clinic. It will help as part of the multiparametric variables to determine the comprehensive risk assessment (estimated 1-year mortality)
Assesment of the right ventricular function by echocardiogram (TAPSE, Right atrial area and pericardial effusion) | 5 years
  Assesment of the right ventricular function by echocardiogram performed by an expert in echocardiography in each scheduled visit (every 6 to 12 months) in the pulmonary hypertension clinic. It will help as part of the multiparametric variables to determine the comprehensive risk assessment (estimated 1-year mortality)
Concentration of serum brain natriuretic peptide | 5 years
  Concentration of serum brain natriuretic peptide in each scheduled visit (every 3 to 6 months) in the pulmonary hypertension clinic. It will help as part of the multiparametric variables to determine the comprehensive risk assessment (estimated 1-year mortality)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Hernandez Oropeza, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No